CLINICAL TRIAL: NCT00894192
Title: Comprehensive Evaluation of Visual Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Chicago Lighthouse (Other)
Collaborators: Ophthonix Inc (Industry); University of Illinois at Chicago (Other)
Responsible Party: Janet Szlyk, PhD, The Chicago Lighthouse
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPH-2005-0516
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Visual Function
Keywords: This study tests functional ability of patients with refractive error or normal vision while using different types of eyeglasses.

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wavefront guided lenses (Active Comparator)
  Interventions: Device: Izon Wavefront-guided lenses
- Conventional lenses (Placebo Comparator)
  Interventions: Device: Conventional lenses

INTERVENTIONS:
Device: Izon Wavefront-guided lenses — Subjects will use prescribed eyeglasses for one week. Their visual functioning will be tested at the end of the week.
  Arms: Wavefront guided lenses
Device: Conventional lenses — We will test the subjects with these lenses after they have worn them for one week. Same procedures will be followed as with the other lenses.
  Arms: Conventional lenses

SUMMARY:
The purpose of this study is to assess the level of visual functioning in patients with various eye conditions while wearing different types of eyeglasses.

DETAILED DESCRIPTION:
The purpose of the research is to study the level of visual functioning in individuals with various eye conditions when using different types of eyeglass lenses. Therefore, the goal of this study is to determine factors that may account for variability in the visual functioning of individuals with a range of refractive errors and their ability to perform everyday activities when equipped with different types of lenses. We hypothesize that the subjects will perform visual tasks of function better when using iZon™ Wavefront-Guided Glasses than with conventional glasses. This hypothesis is based upon the glasses yielding better visual acuity and because the design of the glasses reduces the effects of glare. This research is important so that alternate treatments and vision correction may be implemented which will have a more beneficial impact on those with refractive errors and visual impairment.

ELIGIBILITY:
Inclusion Criteria:

* Have normal vision
* Are far-sighted or near-sighted
* Have no eye diseases Subjects aged 18 and over, who have refractive errors ranging from +5.0 to -5.0 and/or who have eye disease will be included in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity, and Contrast Sensitivity | Once a week

CONTACTS AND LOCATIONS:
Locations (1):
- The Chicago Lighthouse, Chicago, Illinois, United States